CLINICAL TRIAL: NCT05190198
Title: Effect of Ankle Proprioception Training in Improving the Balance in Patients of Type 2 Diabetic Neuropathy
Brief Title: Effect of Ankle Proprioception Training in Type 2 Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00819 Anam
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive ankle proprioceptive training.
  Ankle proprioceptive training includes the following group of exercises:
  1. Training on the floor for 10 minutes (1-8 weeks)
  2. Training on balance pad for 10 minutes (1-4 weeks)
  3. Training on rocked balance board for 10 minutes (5-8 week)
  Interventions: Other: Proprioceptive neuromuscular facilitation
- Conventional therapy group (Active Comparator): The control group will receive Traditional physical therapy exercises.
  1. Active range of motion exercises for ankle and subtalar joints for 5 minutes.
  2. Functional balance training for 15 minutes involving
  3. Gait training for 10 minutes.
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: Proprioceptive neuromuscular facilitation — * Weight shifting in each direction (anteriorly, posteriorly, and lateral side) combined with side-to-side head movements (5 times for each direction).
  * One-legged stance with slight knee flexion of another leg for 15 seconds (5 times for each leg).
  * One-legged stance with increasing knee flexion of the other leg for 15 seconds (5 times for each leg).
  * Standing on a balance pad with shifting weight (anteriorly, posteriorly, and lateral side) 10 times in each direction.
  * In standing position, moving the weight left and right maximally.
  * In standing position, moving the weight forward and backward maximally.
  * In standing position, moving both heels of feet up and down.
  * In standing position, bending and stretching both knees by squatting as much as possible.
  Arms: Experimental group
Other: conventional therapy — (Dorsiflexion, planter flexion, eversion and inversion) 10 repetitions for each movement.
  (A) Sit to stand (5 times). (B) Standing with shifting Weight anteriorly, posteriorly, and sideway (5 times for each direction). (C) Functional reach sideway and anterior for touching targets set by the therapist (5 times for each direction). (D) Standing on heels for 20 seconds (5 times). (E) Standing on toes for 20 seconds (5 times).
  (A) Spot marching (2 min). (B) Walking over the heels, toes, lateral border of feet with the preferred speed (6 min). (C) Tandem walking in a straight line (2 min).
  Arms: Conventional therapy group

SUMMARY:
Diabetes mellitus is a metabolic disease described by hyperglycemia, which results from deficiencies in insulin secretion, the action of insulin on the target tissue, both. Chronic hyperglycemia can lead to long-standing damage and failure of various organs, including the kidneys, heart, eyes, blood vessels, and nerves. Diabetes mellitus is one of the world's biggest public health problems, affecting about 415 million people worldwide among adults aged 20 to 79 years. Patients with type 2 diabetic neuropathy (DN) are at increased risk of falls. This increased risk is likely because of the well-documented balance problems attributed to neuropathy and sensory ataxia, which is the lack of precise proprioceptive feedback. Sources of instability in patients with type 2 DN include loss or reduction of peripheral sensory information in the feet, the inability of the central nervous system (CNS) to appropriately integrate the available postural control information, and the shift from an ankle-based method to a hip-based balance strategy. In addition, increased use of vestibular information and reliance on visual information alter the style of postural control in patients with diabetic neuropathy. Individuals with diabetic peripheral neuropathy (DPN) are 15 times more likely to experience falls compared to healthy subjects.

DETAILED DESCRIPTION:
Proprioception can help with joint stability, postural control, and many other conscious sensations. The diabetes mellitus patients showed a decrease in the reflex responses to postural disturbance followed by a decrease in the speed of nerve conduction which leads to disturbance of the balance and increases the risk of falls.The hip and ankle joints play important roles in the control of balance.The major functions of the ankle joint are control of balance against postural disturbances, shock absorption during walking, and movement of the lower limbs. To provide these, it is necessary to maintain a sufficient range of motion of the ankle joint, muscle strength, and proprioceptive sense.

A study reported that both proprioception exercise training and backward walking training are effective in increasing the proprioception sensation of lower limbs. However, proprioception exercise training was better than backward walking training in improving the feeling of proprioception in the lower limbs of patients with diabetic neuropathy. a study was conducted to investigate the effectiveness of an ankle proprioceptive control program on the gait of patients with chronic stroke. The study results provide evidence to support the effectiveness of an ankle proprioceptive control program in improving gait ability of patients with chronic stroke. A study reported that the addition of ankle proprioceptive training to traditional physical therapy exercises could provide more improvement of gait ability and decrease the risk of falling in patients with diabetic neuropathy.

Proper evidence behind ankle proprioception training in the improvement of balance in diabetic neuropathy patients is sparse and is based on different clinical experiences and fewer studies with limited methodological design. Despite the strong relationship between ankle proprioception and gait ability which has been reported in the previous research studies, up till now, there is no study to assess to what extent ankle proprioceptive training can improve balance in patients with diabetic neuropathy. So, the current study will investigate the effects of ankle proprioceptive training in improving the balance in patients with diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients having peripheral neuropathy previously diagnosed by physician / Modified Toronto Clinical Neuropathy Score 9-11 = moderate neuropathy; ≥ 12 = severe neuropathy
* Type II diabetes mellitus
* Timed up and go test <20 sec
* Berg Balance score between 20-40
* Able to walk without assistance or assistive device
* controlled blood glucose level

Exclusion Criteria:

* Cognitive Deficits
* Severe retinopathy
* Severe nephropathy that causes edema or needs hemodialysis.
* Scars under their feet
* Other neurological or orthopedic impairments (such as stroke, poliomyelitis, rheumatoid arthritis, or severe osteoarthritis)
* Any medical conditions that would confound the assessment of neuropathy, such as malignancy, active/untreated thyroid disease.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Fall Efficiency Scale-International (FES-I) | week 8
  Risk of falling is assessed with Fall Efficiency Scale- International (FES-I). This is a self-reported 16-item scale of perceived confidence to complete physical daily activities. It scored each item on a four-point scale (1 = not at all concerned, 2 = somewhat concerned, 3 = fairly concerned and 4 = very concerned). The possible total score is 64 in the worst case and 16 in the best condition to do all tasks with no concern of falling.
Timed up and go test (TUG) | week 8
  The Timed Up and Go (TUG) is a screening tool used to test basic mobility skills of frail elderly patients (60-90 years old). They can use the TUG with but is not limited to, persons with stroke.
  10s Completely independent With or without walking aid for ambulation and transfers
  < 20s Independent for main transfers With or without walking aid, independent for basic tub or shower transfers and able to climb most stairs and go outside alone
  > 30s Requires assistance dependent in most activities
Berg Balance Scale | week 8
  The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item comprising a five-point ordinal scale ranging from 0 to 4, with 0 showing the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete.
Modified Toronto Clinical Neuropathy Score (mTCNS) | week 8
  It is a screening tool for diabetic peripheral neuropathy and correlates with the severity of diabetic neuropathy. The mTCNS comprises two sub-scores only: symptom score and sensory test score. The values of the symptoms score range between 0 and 18 points.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Afridi, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Maryam Day Care Clinic Kallar Kahar, Kallar Kahar, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atre JJ, Ganvir SS. Effect of functional strength training versus proprioceptive neuromuscular facilitation on balance and gait in patients with diabetic neuropathy. Indian Journal of Physical Therapy and Research. 2020;2(1):47
- [Background] Ahmad I, Hussain E, Singla D, Verma S, Ali K. Balance training in diabetic peripheral neuropathy: A Narrative Review. JSM Diabetol Manag. 2017;2(1):1002.
- [Background] Dominguez-Muñoz FJ, Hernández-Mocholi MA, Manso LJ, Collado-Mateo D, Villafaina S, Adsuar JC, et al. Test-retest reliability of kinematic parameters of timed up and go in people with type 2 diabetes. Applied Sciences. 2019;9(21):4709.
- [Background] Skamagas M, Breen TL, LeRoith D. Update on diabetes mellitus: prevention, treatment, and association with oral diseases. Oral Dis. 2008 Mar;14(2):105-14. doi: 10.1111/j.1601-0825.2007.01425.x. PMID 18302671
- [Background] Olokoba AB, Obateru OA, Olokoba LB. Type 2 diabetes mellitus: a review of current trends. Oman Med J. 2012 Jul;27(4):269-73. doi: 10.5001/omj.2012.68. PMID 23071876
- [Background] Khan MAB, Hashim MJ, King JK, Govender RD, Mustafa H, Al Kaabi J. Epidemiology of Type 2 Diabetes - Global Burden of Disease and Forecasted Trends. J Epidemiol Glob Health. 2020 Mar;10(1):107-111. doi: 10.2991/jegh.k.191028.001. PMID 32175717
- [Background] Asiimwe D, Mauti GO, Kiconco R. Prevalence and risk factors associated with type 2 diabetes in elderly patients aged 45-80 years at Kanungu District. Journal of diabetes research. 2020;2020.
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2014 Jan;37 Suppl 1:S81-90. doi: 10.2337/dc14-S081. No abstract available. PMID 24357215
- [Background] Saleh MS, Rehab NI. Effect of ankle proprioceptive training on gait and risk of fall in patients with diabetic neuropathy: A randomized controlled trial. International Journal of Diabetes Research. 2019;2(1):40-5.
- [Background] Jeannin AC, Salem JE, Massy Z, Aubert CE, Vermeer C, Amouyal C, Phan F, Halbron M, Funck-Brentano C, Hartemann A, Bourron O. Inactive matrix gla protein plasma levels are associated with peripheral neuropathy in Type 2 diabetes. PLoS One. 2020 Feb 24;15(2):e0229145. doi: 10.1371/journal.pone.0229145. eCollection 2020. PMID 32092076